CLINICAL TRIAL: NCT01522469
Title: A Phase II Study of Crenolanib Besylate in Subjects With Relapsed/Refractory Acute Myeloid Leukemia With FLT3 Activating Mutations
Brief Title: Phase II Study of Crenolanib in Subjects With Relapsed/Refractory AML With FLT3 Activating Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-004
Record Dates: First submitted 2012-01-30; First posted 2012-01-31 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia With FLT3 Activating Mutations
Keywords: FLT3; Crenolanib; Acute; myeloid; leukemia; relapsed; refractory
MeSH Terms: conditions — Recurrence; Leukemia

ARMS (1):
- Crenolanib Besylate (Experimental)
  Interventions: Drug: Crenolanib Besylate (CP-868,596-26)

INTERVENTIONS:
Drug: Crenolanib Besylate (CP-868,596-26) — Subjects will take crenolanib 200mg/m2/day divided in three doses daily (preferably every eight hours), taken orally at least 30 minutes pre or post meal until disease progression, death, or the patient discontinues treatment for adverse events, investigator's judgment, or other reasons. Patients who are able to proceed to allogeneic stem cell transplant will be able to resume crenolanib therapy post-transplant in an attempt to maintain remission.

SUMMARY:
This is a Phase II open label study of crenolanib besylate. This study will enroll subjects with relapsed or refractory AML with FLT3 activating mutations. Prior treatment with other FLT3 TKIs is allowed. Subjects will take crenolanib 200mg/m2/day divided in three doses daily (preferably every eight hours), taken orally at least 30 minutes pre or post meal until disease progression, death, or the patient discontinues treatment for adverse events, investigator's judgment, or other reasons. Patients who are able to proceed to allogeneic stem cell transplant will be able to resume crenolanib therapy post-transplant in an attempt to maintain remission.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory primary AML or AML secondary to antecedent hematologic disorder with an expected survival of 3 months or greater
* Patients must have tested positive for FLT3-ITD and /or other FLT3 activating mutations within < 60 days of the screening period.
* Age ≥18 years
* ECOG PS 0 - 2
* Adequate liver function, defined as total or direct bilirubin ≤1.5x ULN, ALT ≤3.0x ULN,AST ≤3.0x ULN. Exceptions for ALT and AST restrictions will be made in the setting of documented liver involvement with leukemia
* Adequate renal function, defined as serum creatinine ≤1.5x ULN
* Recovery from non-hematological toxicities of prior therapy (including HSCT) to no more than grade 1 (except alopecia)
* Subjects should have received no anti-leukemic therapy (except hydroxyurea) prior to the first dose of crenolanib as follows: for 14 days for classical cytotoxic agents and for five times the t1/2 (half-life) for FLT3 inhibitors and antineoplastic agents that are neither cytotoxic nor FLT3 inhibitors (e.g. hypomethylating agent or MEK inhibitor)
* Negative pregnancy test for women of childbearing potential
* Able and willing to provide written informed consent
* Subjects who received crenolanib prior to and are within 30-90 days of an allogeneic stem cell transplant (HSCT) and have either no active GVHD where therapy has been initiated or GVHD where therapy has not been escalated within 14 days prior to start of study drug

Exclusion Criteria:

* Absence of FLT3 activating mutation
* <5% blasts in blood or marrow at screening
* Concurrent chemotherapy, systemic immunosuppressants, or targeted anti-cancer agents,other than hydroxyurea
* Patient with concurrent severe and/or uncontrolled medical conditions that in the opinion of the investigator may impair the participation in the study or the evaluation of safety and/or efficacy
* HIV infection or active hepatitis B manifested as hepatitis surface antigen positive (HepBsAg) or hepatitis C manifested as hepatitis C antibody positive
* For post HSCT, subjects who are within 29 days of an allogeneic transplant, and/or are on an unstable dose of immunosuppressive drugs for management or prophylaxis of GVHD or have escalated therapy for GVHD within 14 days of starting study drug and/or have >/=Grade 2 persistent non hematological toxicity related to the transplant or did not receive crenolanib prior to HSCT
* Evidence of lack of engraftment if post allogeneic transplant
* Unable to swallow pills
* Major surgical procedures within 14 days of Cycle 1 Day 1 administration of crenolanib
* Unwillingness or inability to comply with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TKI Pre-treated: Participants who had relapsed/refractory AML with FLT3 activating mutations whose leukemia progressed and have a history of prior therapy with one or more FLT3 TKIs received either 200mg/m2 /day crenolanib divided in three doses daily or 100mg TID depending on the version of the protocol at the time of their enrolment. (preferably every eight hours), taken orally at least 30 minutes pre or post meal. Crenolanib was taken orally at the abovementioned doses at least 30 minutes pre or post meal until disease progression, death, or the patient discontinues treatment for adverse events, investigator's judgment, or other reasons. Patients who were able to proceed to allogeneic stem cell transplant were able to resume crenolanib therapy post-transplant in an attempt to maintain remission.
- TKI Naive: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one or more prior chemotherapy regimens excluding any FLT3 TKI received either 200mg/m2 /day crenolanib divided in three doses daily or 100mg TID depending on the version of the protocol at the time of their enrolment. (preferably every eight hours), taken orally at least 30 minutes pre or post meal. Crenolanib was taken orally at the abovementioned doses at least 30 minutes pre or post meal until disease progression, death, or the patient discontinues treatment for adverse events, investigator's judgment, or other reasons. Patients who were able to proceed to allogeneic stem cell transplant were able to resume crenolanib therapy post-transplant in an attempt to maintain remission.
Period: Overall Study
Arm/Group | TKI Pre-treated | TKI Naive
Started | 9 | 4
Completed | 9 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TKI Pre-treated | TKI Naive | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 4 | 1 | 5
  45 to 60 years | 3 | 1 | 4
  Greater than 60 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  White | 8 | 4 | 12
FLT3 status [Count of Participants; unit: Participants] — Mutations in the gene encoding the trans-membrane tyrosine kinase FLT3. The type of FLT3 mutation detected by bone marrow assessment at diagnosis was collected. Subjects had either internal tandem duplications (ITD) in the juxtamembrane domain, point mutations or deletions in the tyrosine kinase domain (TKD) or both ITD and TKD mutations together.
  Participants
    FLT3-ITD | 1 | 2 | 3
    FLT3-D835 | 0 | 0 | 0
    FLT3-ITD and D835 | 8 | 2 | 10
Number of prior therapies [Median (Full Range); unit: number of lines of therapy] | 3 [2 to 6] | 1.5 [1 to 3] | 2 [1 to 6]
Baseline ECOG Performance [Count of Participants; unit: Participants] — ECOG performance status graded by the investigator during a physical assessment. A greater ECOG grade is associated with greater impact of the disease on the ability of the subject to live. Grade 0 indicates subjects who are fully active and able to carry on all pre-disease performance. Grade 1 indicates subjects restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. Grade 2 indicates subjects who are ambulatory and capable of all selfcare but unable to carry out any work activities.
  Participants
    ECOG 0 | 0 | 1 | 1
    ECOG 1 | 6 | 3 | 9
    ECOG 2 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the response rate to crenolanib.Complete remission (CR) response criteria include a post-baseline bone marrow (BM) biopsy or aspiration % blasts <5%, absolute neutrophil count (ANC) >1×10^9/L and platelet count >100×10^9/L. CRi response included all CR criteria met, except participant did not experience either platelet recovery or ANC recovery. Partial Response (PR) response included a decrease of ≥50% in % blasts in the BM aspirate or biopsy from baseline but >5%. Hematologic improvement (HI) response included erythroid response where Hgb increased ≥ 1.5 g/dL, platelet response where platelets increased ≥ 30 x 10^9/L for patient starting with >20 x 10^9/L platelets or increase from <20 x 10^9/L to >20 x 10^9/L and by at least 100% and neutrophil response where at least 100% increase and an increase >0.5 x 10^9/L. Resistant Disease (RD) was defined as the absence of CR, CRi, CRp, PR or HI.
Time Frame: From the date of first dose to the end of protocol treatment, 1 year.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Participants who had relapsed/refractory AML with FLT3 activating mutations who progressed on one or more prior chemotherapy regimens received either 200mg/m2 /day crenolanib divided in three doses daily or 100mg TID depending on the version of the protocol at the time of their enrolment. (preferably every eight hours), taken orally at least 30 minutes pre or post meal. Crenolanib was taken orally at the abovementioned doses at least 30 minutes pre or post meal until disease progression, death, or the patient discontinues treatment for adverse events, investigator's judgment, or other reasons. Patients who were able to proceed to allogeneic stem cell transplant were able to resume crenolanib therapy post-transplant in an attempt to maintain remission.
Arm/Group | All Patients | TKI Pre-treated | TKI Naive
Number analyzed (Participants) | 13 | 9 | 4
Participants
  CR/CRi | 5 | 2 | 3
  PR | 1 | 1 | 0
  HI | 3 | 2 | 1
  ORR (CR+PR) | 6 | 3 | 3
  Clinical Benefit (CR+PR+HI) | 9 | 5 | 4
  RD | 4 | 4 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30-days after the last dose, 1 year.
Description: Safety data was presented in a comprehensive manner since no formal arms existed as part of the study; patients were only categorized this way during post-study data analyses to determine if there was a potential relationship between their prior TKI exposure and their response to crenolanib therapy.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 13/13
Serious Adverse Events (participants affected / at risk) | 12/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 3
Multiple organ dysfunction syndrome (General disorders) | 2
Multi-organ failure (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pyrexia (General disorders) | 1
Sepsis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Liver function test increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Anemia (Blood and lymphatic system disorders) | 4
Pancytopenia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 3
Cardiomegaly (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Ocular icterus (Eye disorders) | 1
Retinal hemorrhage (Eye disorders) | 1
Vitreous hemorrhage (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 4
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oral mucosal blistering (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Tongue ulceration (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Oedema peripheral (General disorders) | 4
Chest pain (General disorders) | 3
Chills (General disorders) | 3
Disease progression (General disorders) | 3
Face oedema (General disorders) | 3
Multiple organ dysfunction syndrome (General disorders) | 3
Oedema (General disorders) | 3
Pain (General disorders) | 3
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 2
Malaise (General disorders) | 2
Multi-organ disorder (General disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 4
Clostridium difficile infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Alpha hemolytic streptococcal infection (Infections and infestations) | 1
Bacteremia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Respiratory synctial virus infection (Infections and infestations) | 1
Staphlococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Blood phosphorus increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 2
Blood albumin decreased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood urea nitrogen/creatinine ratio (Investigations) | 1
Blood urea nitrogen/creatinine ratio increased (Investigations) | 1
Cardiac murmur (Investigations) | 1
Gamma-glutamyl transferase increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Monocyte count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Abnormal loss of weight (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypervolemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypoproteinemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 2
Hypoesthesia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 2
Hallucination (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Vaginal oedema (Reproductive system and breast disorders) | 1
Vulval disorder (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1
Hair color changes (Skin and subcutaneous tissue disorders) | 1
Madarosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT01522469/Prot_SAP_000.pdf